CLINICAL TRIAL: NCT03898362
Title: Clinical Evaluation of Pneumatic Technology for Powered Mobility Devices
Brief Title: Pneumatic Technology for Powered Mobility Devices
Acronym: PTPMD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19 made completion of clinical trial portion impossible
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A2753-R
Record Dates: First submitted 2019-03-15; First posted 2019-04-02 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Disability
Keywords: wheelchair; scooter

STUDY DESIGN:
Intervention Model Description: 6 months using one device then crossover and 6 months using other device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- pneumatically powered wheelchair or scooter (Active Comparator): participants will use pneumatic powered wheelchair or scooter
  Interventions: Other: pneumatically powered wheelchair or scooter
- battery powered wheelchair or scooter (Active Comparator): participants will use battery powered wheelchair or scooter
  Interventions: Device: battery powered wheelchair or scooter

INTERVENTIONS:
Other: pneumatically powered wheelchair or scooter — a wheelchair or scooter powered by compressed air will be used for 6 months. Compressed air is a novel power source and no batteries are used in these devices.
  Arms: pneumatically powered wheelchair or scooter
Device: battery powered wheelchair or scooter — a wheelchair or scooter powered by a battery will be used for 6 months. These are conventional mobility devices that the participants are using or in the process of obtaining
  Arms: battery powered wheelchair or scooter

SUMMARY:
Over 240,000 Veterans with disabilities use mobility devices such as manual and power wheelchairs and scooters, and this number continues to grow. Mobility devices have been described as the most enabling technology a clinician can provide to a person with a disability. Yet, the batteries used to power scooters and wheelchairs have many drawbacks. Batteries are hazardous to humans and the environment, heavy (which limits transportability), and incompatible with wet or highly humid environments. Repairs to electrical systems and replacement of batteries are frequently needed. These are costly and adversely affect the Veteran. Compressed air is a power source that overcomes many of these disadvantages. The investigators have developed a scooter and a wheelchair that are powered solely by compressed air. The purpose of this study is to clinically evaluate the impact of these new devices on Veterans living in long-term care facilities, and to obtain feedback from nurses, therapists, and engineers regarding their design and feasibility of use in long-term care.

DETAILED DESCRIPTION:
Over 240,000 Veterans with disabilities use mobility devices such as manual and power wheelchairs and scooters, and this number continues to grow. Mobility devices have been described as the most enabling technology a clinician can provide to a person with a disability. Appropriate mobility devices improve function, independence, home and community integration; activity and participation; comfort; and quality of life. Yet, battery-powered mobility devices (BPMDs) have many drawbacks. Despite advances in technology, batteries are still hazardous to humans and the environment, heavy (which limits transportability), and incompatible with wet or highly humid environments. Repairs to electrical systems and replacement of batteries are frequently needed. These are costly and result in being stranded, missing medical appointments, missing work or school, injury, increased pain, lower self-perceived health, skin breakdown, higher hospitalization rates, and reduced community participation. Surveys conducted by the VA Center on Wheelchairs and Associated Rehabilitation Engineering (WARE) identified alternative power sources as a top research priority of Veterans and providers.

Compressed air is a power source that has many advantages over batteries, including safety to both humans and the environment, lighter weight, waterproof nature, and lack of any electrical components which can reduce the frequency of repairs. Two novel pneumatically-powered mobility devices (PPMDs), a scooter and wheelchair, were developed and tested for feasibility with 107 users. The devices were lighter and had sufficient driving range per charge for the average user. There were no safety or repair issues encountered in the 11-week field test. Filling air tanks was also much faster than charging a typical battery. With pilot funds, the investigators then built two new scooters and two new power wheelchairs with longer driving ranges. The investigators also developed a portable backup tank system that allows us to refill or replace the tanks easily in the community.

The purpose of this study is to clinically evaluate the impact of PPMDs on Veterans living in long-term care facilities, and to obtain feedback from key stakeholders regarding the design and feasibility of use of PPMDs in long-term care. Long-term care was chosen because it is an ideal setting for technology that is water-proof (e.g., compatible with inclement weather, ease of cleaning, and resistant to incontinence and requires less maintenance and upkeep. In Phase 1 (Technical), the investigators will build 8 pneumatically-powered scooters, 8 pneumatically-powered wheelchairs, 2 air filling stations with flow switches that measure air filling time, 20 dataloggers that will measure battery charging time, and 20 dataloggers that will monitor activity levels. Phase 2 (clinical evaluation) will comprise two aims. First, the investigators will enroll 50 Veterans into a cross-over trial in which they use a BPMD provided to them that is the same make and model as their own BPMD, and its PPMD counterpart in random order, each for 6 months. The investigators will compare pneumatically-powered and battery-powered scooters and wheelchairs with respect to functional mobility, satisfaction, psychosocial impact, "charging time," maintenance and repairs. The investigators hypothesize that Veterans will have higher levels of mobility, satisfaction, and psychosocial impact when using PPMDs compared to when using BPMDs. The investigators also hypothesize that PPMDs will be faster to "charge" and have fewer maintenance and repair issues than BPMDs. Second, the investigators will conduct qualitative interviews of the 50 participants in the clinical evaluation and an additional 54 key stakeholders involved in PPMD and BPMD use (e.g., family members/caregivers, clinicians, and technical support personnel). The investigators will assess patient, facility, VA healthcare system, and other factors that may be barriers or facilitators to use of PPMDs and identify modifiable factors that may further improve the design.

Results of the proposed study will pave the way for potential adoption of this technology within the VA. Such adoption could have a direct and positive impact on Veterans' lives. This research has the potential for national impact on the wheelchair provision process and services within the VA.

ELIGIBILITY:
Inclusion Criteria:

Aim 2A

* Participant must be 18 years or older
* Participant must use or be in the process of obtaining a scooter or Group 2 power wheelchair without power seat functions
* Participant must be able to speak and understand English in order to provide informed consent

Aim 2B Inclusion Criteria

* Participants must be 18 years or older
* Participants must be either a participant in Aim 2A, a family member/caregiver of a participant, or an employee of a participating long-term care facility
* Participants who are employees must have some experience with charging, storing, transporting, cleaning, or maintaining BPMDs, e.g.:

  * nurse
  * physical therapist
  * occupational therapist
  * engineer, etc.
* Participants who are employees must be willing to assist at least three Aim 1 participants in the charging, storing, transporting, cleaning, or maintaining of their PPMDs for at least 3 months
* Participants must be able to speak and understand English in order to provide informed consent

Exclusion Criteria:

Exclusion Criteria for Aim 2A

* Open pressure injuries of skin on sitting surface that could worsen with prolonged sitting

Exclusion Criteria for Aim 2B

* There are no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad E. Dicianno, MD MS, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were randomized into the cross-over sequences and the planned cross-over study was not conducted
Groups:
- Expert: healthcare professional
- Veteran With Disability: Veteran with disability who has experience using wheelchairs or scooters
Period: Overall Study
Arm/Group | Expert | Veteran With Disability
Started | 14 | 6
Completed | 14 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Veterans With Disability: Veterans with disability with experience using wheelchairs and scooters
- Total: Total of all reporting groups
Arm/Group | Expert | Veterans With Disability | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (10.3) | 70.4 (3.3) | 52.3 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 13 | 5 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 12 | 2 | 14
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 6 | 20
Number of people with spinal cord injury [Number; unit: participants] | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Mobility Assessment
Description: Functional measure of mobility; change of 10 points is considered clinically significant. The FMA contains 10 items that measure the extent to which a mobility device aids a user in completing functional tasks like reaching, personal care tasks, indoor mobility, outdoor mobility and transferring. Ten items are scored individually on a 7- point Likert scale (6 = completely agree, 5 = mostly agree, 4 = slightly agree, 3 = slightly disagree, 2 = mostly disagree, 1 = completely disagree and 0 = does not apply to me). A total mobility score is then calculated from summing the individual item scores and an adjusted total score is expressed as a percentage of total score divided by sum of relevant items. The FMA is the most widely used measure to assess function in mobility device users. The change in FMA will be assessed 3 times over a 6 month period in each arm of the trial. Assessments will occur in month 1, 3 and 6 within the first 6 months and repeated in the second 6 months.
Time Frame: Month 1, 3 and 6 within the first 6 months and repeated in the second 6 months.
Population: This outcome measure could not be conducted, and data were not collected due to COVID-19
Arm/Group | Expert | Veteran With Disability
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline
Description: The clinical trial did not occur because of COVID-19
Arm/Group | Expert | Veteran With Disability
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6
Other Adverse Events (participants affected / at risk) | 0/14 | 0/6

LIMITATIONS AND CAVEATS:
No participants were randomized into the cross-over sequences and the planned cross-over study was not conducted because of COVID-19. All participants reported participated in one focus group. Each participant's duration of participation was one day, and no adverse events occurred during the day of their participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-07-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT03898362/Prot_001.pdf
  • Statistical Analysis Plan (2025-07-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT03898362/SAP_002.pdf
  • Informed Consent Form (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT03898362/ICF_000.pdf